CLINICAL TRIAL: NCT07332780
Title: A Randomized Controlled Study of Adenotonsillectomy on Spinal Curve Magnitude in Children With Mild Sleep-Disordered Breathing
Brief Title: Effect of Adenotonsillectomy on Spinal Curve Magnitude in Children With Sleep-Disordered Breathing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Ningbo No. 1 Hospital (Other); Ningbo No.2 Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Xiangyang Wang, M.D., Chief physician, Doctorial supervisor, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHWenzhouMU-CR2025K-261-01
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sleep-disordered Breathing (SDB); Idiopathic Scoliosis; Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive | interventions — Adenoidectomy; Watchful Waiting; Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologists measuring Cobb angles will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Adenotonsillectomy (eAT) surgery (Active Comparator): There will be removal of tonsils and adenoids that will be performed within 4 weeks of the baseline visit.
  Interventions: Procedure: Adenotonsillectomy (AT) - removal of adenoids and tonsils
- Watchful Waiting with Supportive Care (WWSC) (Other): Children will be closely monitored and re-evaluated for AT by an otolaryngologist after the primary 12 month monitoring period.
  Interventions: Other: Watchful Waiting with Supportive Care

INTERVENTIONS:
Procedure: Adenotonsillectomy (AT) - removal of adenoids and tonsils — Standard clinical adenotonsillectomy within 4 weeks post randomization in addition to information about healthy sleep habits for children and appropriate clinical referrals for management of co-morbidities.
  Arms: Early Adenotonsillectomy (eAT) surgery
Other: Watchful Waiting with Supportive Care — Children will receive information about healthy sleep habits and appropriate clinical referrals for management of co-morbidities. They will be closely monitored and re-evaluated for AT after the primary 12 month monitoring period.
  Arms: Watchful Waiting with Supportive Care (WWSC)

SUMMARY:
This study aims to determine the effect of adenotonsillectomy (AT) surgery on the progression of spinal curvature in children with mild sleep-disordered breathing (SDB) and concurrent scoliosis, as well as its potential role in preventing the de novo development of scoliosis in children with SDB.

DETAILED DESCRIPTION:
Idiopathic scoliosis (IS) is the most common spinal deformity and is frequently associated with abnormal respiratory function. Despite extensive research, its etiology remains unclear, lacking modifiable targets for prevention or early intervention. Notably, studies report a high prevalence of obstructive sleep apnea (OSA) in adolescents with IS (approximately 19.8%-32.9%), and the incidence of SDB symptoms like snoring and OSA can be as high as 42.7% in children with early-onset scoliosis, often leading to ENT referrals for AT. While SDB is known to adversely affect child development, behavior, and cognition, it remains unclear whether this prevalent condition also influences the onset and progression of scoliosis. If so, prolonged exposure to SDB may exert a sustained impact on spinal alignment, potentially persisting even after the causative factor is removed. Therefore, evaluating the effect of SDB and its elimination on spinal curvature is warranted.

Adenotonsillectomy is a first-line treatment for pediatric SDB and one of the most common surgeries performed under general anesthesia in children, proven to resolve SDB in most cases. A recent small retrospective study reported a high rate of scoliosis in children with SDB and a general reduction in Cobb angle post-AT, particularly in younger children, suggesting SDB may be a modifiable target in IS. We hypothesize that SDB and associated intermittent hypoxia due to adenotonsillar hypertrophy increase the risk of de novo and progressive IS, and that spinal curvature will change following AT in children with SDB.

This prospective, single-blind, randomized controlled trial will be conducted at the "Pediatric SDB-Spine Health" Center. All subjects will be diagnosed with SDB via sleep questionnaire (PSQ), ENT examination, and overnight laboratory polysomnography (PSG). Concurrently, all SDB subjects will undergo standard scoliosis screening; those with a Cobb angle ≥ 10° on baseline X-ray will be diagnosed with scoliosis. Following the design of landmark trials like CHAT and PATS, eligible children will be randomized into two groups. One group will undergo early AT within one month of enrollment, while the other will enter a Watchful Waiting with Supportive Care (WWSC) group, with surgical re-evaluation scheduled at ≥12 months post-enrollment. Routine follow-up visits will be scheduled at 6-month intervals for at least 24 months to assess curve progression in children with pre-existing scoliosis. Children with SDB but without scoliosis at baseline will also undergo annual scoliosis screening as part of an ongoing Zhejiang provincial health initiative. Given the high individual prevalence of both SDB and scoliosis in the pediatric population, this study holds significant public health importance.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 15 years.
2. Diagnosed with mild SDB, defined as: Obstructive Apnea-Hypopnea Index (OAHI) ≤5 events/hour on a laboratory-based PSG performed within the past 6 months, AND parental report of habitual obstructive breathing symptoms (e.g., snoring, mouth-breathing, witnessed apneas) occurring >3 nights per week on average.
3. Tonsillar hypertrophy grade ≥2 (on a scale of 0-4) and deemed an appropriate candidate for AT upon ENT evaluation (i.e., no absolute contraindications such as submucous cleft palate).
4. Has undergone radiographic screening for idiopathic scoliosis at the first clinic visit.
5. Skeletally immature (Risser sign 0-3) with spinal Cobb angle < 40 degrees.
6. Informed consent/assent provided by the participant and guardian.

Exclusion Criteria:

1. Unwillingness or inability to comply with study procedures.
2. Plans to relocate outside the study area within 24 months.
3. Previous tonsillectomy or adenoidectomy.
4. Recurrent tonsillitis meeting guideline criteria for immediate AT.
5. Severe OSA (OAHI >10 or as per clinician judgment) or significant hypoxemia requiring immediate CPAP therapy.
6. Severe chronic conditions that could confound outcomes, including but not limited to:

   * Known syndromic, neuromuscular, or congenital musculoskeletal causes of scoliosis.
   * History of spine surgery or significant spinal injury.
   * Spinal tumor.
   * Leg length discrepancy >20 mm.
   * Severe cardiopulmonary disease (e.g., cystic fibrosis, congenital heart disease).
   * Significant cardiac arrhythmia noted on PSG.
   * Bleeding disorders, Sickle Cell Disease.
   * Uncontrolled diabetes, narcolepsy, or asthma.
   * Known genetic, craniofacial, neurological, or psychiatric conditions likely to affect the airway or study participation.
   * Severe obesity (BMI z-score ≥ 3).

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Scoliosis Curve Angle | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  A long standard standing whole spine radiograph will be used for measuring curve size in terms of Cobb angle according to the standard Cobb method
Angle of Trunk Rotation | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  In addition to spinal X-rays, a Scoliometer can also help monitor curve progression. The Scoliometer is an inclinometer that measures the asymmetries between the sides of the trunk by measuring axial rotation in degrees. Numerous studies have found a high correlation between trunk axial rotation (ATR) values and the Cobb angles.

SECONDARY OUTCOMES:
Scoliosis Research Society-22 (SRS-22) questionnaire | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  The SRS-22 aims to evaluate health-related quality of life (HRQOL) in patients with idiopathic scoliosis. The SRS-22 specifically addresses areas affected by spinal deformities-such as pain, self-perception, function, mental health, and satisfaction with treatment. Consequently, it offers a focused approach to understanding the patient experience.
Sleep Measurements | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  Sleep questionnaire with or without further PSG evaluation
Circadian rhythm Measurements | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  Circadian rhythm as assessed by Morning and Evening Questionnaire-5 (MEQ-5)
Body mass index | Routine follow-up visits will be scheduled 6 months apart up to 24 months
  Changes in height, weight and body mass index
Change in Serum Concentration of biomarkers | At baseline and months 12
  Change in serum concentration of Inflammatory Cytokines (IL-6, TNF-α) / Bone Metabolism Markers (PINP) / Oxidative Stress Markers as measured by enzyme-linked immunosorbent assay (ELISA).
Change in Gene Expression Levels of biomarkers | At baseline and months 12
  Change in mRNA expression levels of specific Genes such as HIF1A, Bmal1 and IGFBPs in peripheral blood mononuclear cells (PBMCs) as measured by quantitative reverse transcription polymerase chain reaction (qRT-PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University,, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided